CLINICAL TRIAL: NCT05438186
Title: A Retrospective, Multi-centre, Non-interventional Study Investigating the Clinical Parameters Associated With Saxenda® Use and Discontinuation in Patients in Turkey. INSPIRE Turkey (INvestigate the Impact of Saxenda® on Patient's Weight In a REal World Setting in Turkey) Study
Brief Title: INSPIRE Turkey :A Research Study Looking at the Clinical Parameters Associated With Use and Discontinuation of Saxenda® in Local Clinical Practice in Turkey by Analysing Past Patient Medical Records
Acronym: INSPIRE Turkey
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled since study start.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4805; U1111-1259-8749 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liraglutide: Participants with obesity who received initial prescription of Saxenda® (liragltuide 3.0 milligrams (mg) once daily) and maintained treatment with Saxenda® for at least 16 weeks, without treatment break, following the initial prescription for weight management.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Participants with obesity who received initial prescription of Saxenda® (liragltuide 3.0 milligrams (mg) once daily)) and maintained treatment with Saxenda® for at least 16 weeks, without treatment break, following the initial prescription for weight management.

SUMMARY:
The study is investigating the use of Saxenda (liragltuide 3.0 milligrams (mg) once daily) for weight management. The primary objective is to investigate the change in body weight after initiation and use of Saxenda ® according to local clinical practice for weight management, on adult participant's in a real world setting in Turkey. The study will last for about 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed consent before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Patients who have polyclinic visits between 01 June 2022 and 31 October 2022 and who have received initial prescription of Saxenda® for weight management at least 52 weeks prior to study enrolment.
* Patients who have maintained treatment with Saxenda® for at least 16 weeks, without treatment break, following the initial prescription.
* Patients who have 12-month follow-up data, even if discontinued Saxenda ® treatment.
* Patients who have body weight measurement at baseline and at least 1 more body weight measurement following the Saxenda® prescription
* Age greater than or equal 18 years at the time of signing informed consent

Exclusion criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patient charts lacking any follow-up information for at least 16 weeks.
* Patients who have been treated with anti-obesity medication for last 12 weeks prior to initiation of Saxenda® treatment.
* Patients who receive GLP-1 receptor agonist for treatment of Type 2 diabetes.
* Patients who have undergone bariatric surgery or use of minimal-invasive weight loss devices (i.e. intragastric balloons, lap bands) within 1 year before starting Saxenda® treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with obesity who received initial prescription of Saxenda® and maintained treatment with Saxenda® for at least 16 weeks, without treatment break, following the initial prescription for weight management.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | At 52th week after treatment initiation
  Measured in Percentage (%).

SECONDARY OUTCOMES:
Percentage of relative change in body weight | At 16th week after treatment initiation
  Measured in % of weight.
Percentage of relative change in body weight | At 26th week after treatment initiation
  Measured in % of weight.
Absolute body weight change | At 16th week after treatment initiation
  Measured in kg.
Absolute body weight change | At 26th week after treatment initiation
  Measured in kg.
Absolute body weight change | At 52th week after treatment initiation
  Measured in kg.
Achievement of greater than or equal to 5% weight loss | At 52th week after treatment initiation
  Measured as Count of participants.
Achievement of greater than or equal to 10% weight loss | At 52th week after treatment initiation
  Measured as Count of participants.
Achievement of greater than or equal to 5% and greater than or equal to 10% weight loss | At 26th week after treatment initiation
  Measured as Count of participants.
Mean dose of Saxenda® | At 16th week after treatment initiation
  Measured in mg/day.
Mean dose of Saxenda® | At 26th week after treatment initiation
  Measured in mg/day.
Mean dose of Saxenda® | At 52nd week after treatment initiation
  Measured in mg/day.
Participants who have discontinued Saxenda® | At 16th week after treatment initiation
  Measured in % of total participants.
Participants who have discontinued Saxenda® | At 26th week after treatment initiation
  Measured in % of total participants.
Participants who have discontinued Saxenda® | At 52nd week after treatment initiation
  Measured in % of total participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com